CLINICAL TRIAL: NCT06458439
Title: Phase IIa Trial to Evaluate Epcoritamab Administered Before and After CAR-T Cell Therapy in Patients With Relapsed or Refractory Large B-cell Lymphomas
Brief Title: Epcoritamab-CAR T Cells for Large B-cell Lymphomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 03424; IRB#855865 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma, Non-Hodgkin; Relapsed Diffuse Large B Cell Lymphoma; Refractory Diffuse Large B-cell Lymphoma; High-grade B-cell Lymphoma; Transformed Indolent Non-Hodgkin Lymphoma to Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epcoritamab (Experimental): Study participants will bridging epcoritamab on Cycles 1-3, Days 1, 8, 15, and 22 (once weekly).
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — * C1D1: fixed priming dose of 0.16 mg subcutaneous injection
  * C1D8: fixed intermediate dose of 0.8 mg subcutaneous injection
  * C1D15 onward: fixed full dose of 48 mg subcutaneous injection
  Other Names: GEN3013; DuoBody -CD3xCD20

SUMMARY:
This study investigates the feasibility and efficacy of epcoritamab treatment before CAR T cells. This study also investigates if, when patients have residual lymphoma after CAR T cells, epcoritamab can help to effectively treat that lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Subject must be able and willing to provide informed consent. In the case where the patient is incapacitated or not otherwise capable, a legally authorized representative (or decision maker when there is not an advanced directive in place) must be willing to provide informed consent on behalf of the patient.
* Able to comply with the study protocol, in the investigator's judgment
* ECOG PS of 0 - 2
* Pathology report confirming eligible diagnosis
* Documented CD20+ tumor cells on most recent biopsy
* Patients will have failed to respond to frontline standard of care therapy containing an anthracycline and anti-CD20 antibody
* Patients will be eligible and consent to be treated with a "commercially available" anti-CD19, 4-1BB, CD3zeta CAR-T cell therapy or anti-CD19, CD28, CD3zeta CAR T cell therapy (for example, tisagenlecleucel, lisocabtagene maraleucel, or axicabtagene maraleucel)
* Patients must have a PET/CT scan (preferred), diagnostic CT scan, or MRI with at least one bi-dimensionally measurable lesion (≥ 1.5 cm for nodal lesions or ≥ 1cm for extra-nodal lesions in largest dimension by low-dose computerized tomography [CT] scan with FDG-uptake ≥ liver)
* Adequate laboratory studies
* Resolution of toxicities from prior therapy to a grade that does not contraindicate trial participation in the opinion of the investigator
* Ability and willingness to take proper contraceptive precautions

Exclusion Criteria:

* Inability or unwillingness of the patient or legally authorized representative (or decision-maker when there is not an advanced directive in place) to provide informed consent.
* Prior solid organ transplantation
* Primary central nervous system (CNS) lymphoma or active secondary CNS involvement by lymphoma at screening as confirmed by magnetic resonance imaging (MRI)/computed tomography (CT) scan (brain) or, if clinically indicated, by lumbar puncture.
* History of autoimmune disease or other diseases resulting in permanent immunosuppression or requiring chronic immunosuppressive therapy (see Exclusion Criteria 5a), with the following exceptions:

  1. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone
  2. Patients with a history of lymphoma-related immune thrombocytopenic purpura or autoimmune hemolytic anemia in remission may be eligible for this study if approved by the Regulatory Sponsor and Principal Investigator
  3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

  i. Rash must cover < 10% of body surface area ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroid iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or corticosteroids (> 20 mg/day prednisone or equivalent for > 2 weeks) within the previous 3 months d. rheumatoid arthritis or similar autoimmune/rheumatic conditions
* Systemic immunosuppressive medications (including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents). However, the following are permitted:

  1. If receiving glucocorticoid treatment at screening, must be a maximum daily dose of prednisone 10 mg (or equivalent) and a total of no more than 140 mg over the last 14 days prior to the first dose of epcoritamab, unless for disease control.
  2. Patients who received a single dose of a systemic immunosuppressant medications (e.g., single dose of dexamethasone for nausea or B symptoms) may be enrolled
  3. The use of inhaled corticosteroids is permitted
  4. The use of mineralocorticoids for management of orthostatic hypotension is permitted
  5. The use of physiologic doses of corticosteroids (< 20 mg/day of prednisone or equivalent) for uses such as management of adrenal insufficiency is permitted
* Known past or current malignancy, other than inclusion diagnoses, except for:

  1. Cervical carcinoma of Stage 1B or less.
  2. Adequately resected, non-metastatic basal cell or squamous cell skin carcinoma.
  3. Non-invasive, superficial bladder cancer.
  4. Prostate cancer with a current PSA level <0.1 ng/mL.
  5. Patients with a malignancy that has been treated with curative intent will also be enrolled if that malignancy is in remission prior to first dose of epcoritamab
* Known clinically significant cardiovascular disease
* Patients with the following active infection(s) could have increased risks for toxicity if treated with bispecific antibody therapy, thus patient will be excluded if:

  1. Positive serologic or PCR test results for acute or chronic HBV infection. Patients whose HBV infection status cannot be determined by serologic test results (www.cdc.gov/hepatitis/hbv/pdfs/serologicchartv8.pdf) must be negative for HBV by PCR to be eligible for study participation. Patients with a history of hepatitis B who are negative for HBV by PCR, will not be excluded but will be placed on suppressive antiviral therapy
  2. Acute or chronic HCV infection. Patients who are positive for HCV antibody must be negative for HCV by PCR to be eligible for study participation. Patients with a history of hepatitis C who have been adequately treated (negative PCR) will not be excluded.
  3. Positive serologic or RT-PCR test results for HIV infection.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major documented infection requiring treatment with IV antibiotics or hospitalization within 2 weeks of enrollment. Empiric or prophylactic antibiotics administered during neutropenia or neutropenic fever without microbiologic evidence of infection do not exclude patients.
* Clinically significant pulmonary disease (e.g., bronchospasm and/or obstructive pulmonary disease) that requires chronic oxygen or corticosteroid use > 20 mg mg/day prednisone or equivalent
* Uncontrolled seizure disorder
* Exposure to live or live attenuated vaccine within 4 weeks prior to signing ICF
* Pregnancy or breast feeding
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of CAR T cell infusion among subjects who receive epcoritamab and undergo leukapheresis | Start of epcoritamab to CAR T-cell infusion
  Whether participants receive CAR T-cell infusion (yes/no)

SECONDARY OUTCOMES:
Incidence and severity of AEs, SAEs from epcoritamab until CAR T cell infusion | Day 1 of epcoritamab until CAR T cell infusion
  Assessment of toxicity via incidence and severity of AEs and SAEs via CTCAE v5
Overall Response Rate after 2 cycles of Epcoritamab | Day 1 of epcoritamab to completion of 2 cycles of epcoritamab
  Percentage of subjects who receive epcoritamab and have a CR or PR by Lugano 2014 criteria prior to CAR T-cells
Incidence and severity of AEs, SAEs after CAR T cell infusion through day 28 visit after CAR T-cell infusion | CAR T cell infusion through day 28 visit after CAR T-cells
  Assessment of toxicity via incidence and severity of AEs and SAEs via CTCAE v5
Day 28 visit response rates post CAR T cell infusion | Day 28 visit after CAR T cell infusion
  Overall response rate as well as complete response rate after CAR T-cells
Progression-free survival, duration of response, and overall survival for those subjects achieving complete response at Day 28 visit post CAR T cell infusion | CAR T cell infusion until last follow-up or death
  Duration of response from day 28 visit after CAR T-cells, progression-free survival and overall survival from CAR T-cell infusion
Incidence and severity of AEs, SAEs from day 28 visit after CAR T-cell infusion until epcoritamab discontinuation | Day 28 visit after CAR T-cell infusion until epcoritamab discontinuation up to 12 cycles of epcoritamab
  Assessment of toxicity via incidence and severity of AEs and SAEs via CTCAE v5
Responses at 3 and 6 months after CAR T-cell infusion for subjects who receive epcoritamab after CAR T-cells | 3 and 6 months after CAR T-cell infusion
  Best overall response rate, overall response rate, and complete response rate at 3 and 6 months after CAR T cell infusion for subjects who receive epcoritamab after CAR T-cells
Duration of response, progression-free survival and overall survival from time of CAR T-cell infusion for subjects who receive post CAR T-cell epcoritamab infusions | From CAR T-cell infusion until date of last follow-up or date of death due to any cause, whichever comes first, assessed up to 5 years from last dose of epcoritamab
  Duration of response from first response after CAR T-cell infusion, progression-free survival and overall survival from CAR T-cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Elise Chong, MD, Principal Investigator — Abramson Cancer Center at the University of Pennsylvania
Locations (1):
- Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No